CLINICAL TRIAL: NCT03597789
Title: The Role of Emotion Regulation and Socialization in Behavioral Parent Training (BPT) Efficiency and Outcomes
Brief Title: Tantrum Tamers 2.0: The Role of Emotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-1040; 1R21MH113887-01A1 (NIH)
Record Dates: First submitted 2018-06-29; First posted 2018-07-24 (Actual); Results first posted 2021-08-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-07

CONDITIONS: Child Behavior; Attention Deficit and Disruptive Behavior Disorders; Problem Behavior
Keywords: Tantrums; Inattentive; Noncompliance
MeSH Terms: conditions — Child Behavior; Attention Deficit and Disruptive Behavior Disorders; Problem Behavior; Patient Compliance

STUDY DESIGN:
Intervention Model Description: All families get the evidence-based treatment, Helping the Noncompliant Child (HNC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Helping the NonCompliant Child Treatment (Other): Families will participate in an average of 8 to 12 weeks of Behavioral Parent Training (BPT), by way of the standard-of-care training program "Helping the Noncompliant Child" (HNC) via weekly sessions and mid-week calls.
  Interventions: Behavioral: Helping the Noncompliant Child (HNC)

INTERVENTIONS:
Behavioral: Helping the Noncompliant Child (HNC) — HNC is a mastery-based, family-focused, clinic-based treatment for young children aged 3-8 years with problem behavior.

SUMMARY:
This study aims to better understand how to best help parents of young children with problem behavior. Problem behaviors vary between and within children, but can include inattention/hyperactivity, tantrums, and/or noncompliance.

DETAILED DESCRIPTION:
If eligible and choose to participate, this study includes:

A baseline assessment which will include asking a series of questions about parent, child and family, as well as parent-child observations.

If eligible for treatment, sessions occur once per week for approximately 8 to 12 weeks. Sessions include new information and lots of practice and discussion about how to make the skills work best for specific families.

After finishing treatment a post-assessment (similar to BL) conducted.

All of the assessments (i.e., video-and audio-recorded), as well as the sessions with a therapist will be recorded (i.e., video recorded).

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant child problem behavior

Exclusion Criteria:

* Current severe symptoms in parent or child that would prohibit participation (e.g., parent current psychotic or substance use disorder)

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Jones, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Department of Psychology & Neuroscience, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB) and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication of primary study results

REFERENCES:
- [Derived] McKee LG, Yang Y, Highlander A, McCall M, Jones DJ. Conceptualizing the Role of Parent and Child Emotion Regulation in the Treatment of Early-Onset Behavior Disorders: Theory, Research, and Future Directions. Clin Child Fam Psychol Rev. 2023 Mar;26(1):272-301. doi: 10.1007/s10567-022-00419-y. Epub 2022 Nov 17. PMID 36385585
- [Derived] Highlander AR, Jones DJ. Integrating Objective and Subjective Social Class to Advance Our Understanding of Externalizing Problem Behavior in Children and Adolescents: A Conceptual Review and Model. Clin Child Fam Psychol Rev. 2022 Jun;25(2):300-315. doi: 10.1007/s10567-021-00369-x. Epub 2021 Sep 17. PMID 34533656
- [Derived] Highlander A, Zachary C, Jenkins K, Loiselle R, McCall M, Youngstrom J, McKee LG, Forehand R, Jones DJ. Clinical Presentation and Treatment of Early-Onset Behavior Disorders: The Role of Parent Emotion Regulation, Emotion Socialization, and Family Income. Behav Modif. 2022 Sep;46(5):1047-1074. doi: 10.1177/01454455211036001. Epub 2021 Aug 11. PMID 34378434
- [Derived] Loiselle R, Parent J, Georgeson AR, Thissen D, Jones DJ, Forehand R. Validation of the Multidimensional Assessment of Parenting: An application of item response theory. Psychol Assess. 2021 Sep;33(9):803-815. doi: 10.1037/pas0001019. Epub 2021 Apr 26. PMID 33900099
- [Derived] Jones DJ, Loiselle R, Zachary C, Georgeson AR, Highlander A, Turner P, Youngstrom JK, Khavjou O, Anton MT, Gonzalez M, Bresland NL, Forehand R. Optimizing Engagement in Behavioral Parent Training: Progress Toward a Technology-Enhanced Treatment Model. Behav Ther. 2021 Mar;52(2):508-521. doi: 10.1016/j.beth.2020.07.001. Epub 2020 Jul 15. PMID 33622517

RESULTS

PARTICIPANT FLOW:
Groups:
- Helping the NonCompliant Child Treatment: Families will participate in approximately 10 weeks of Behavioral Parent Training (BPT), by way of the standard-of-care training program "Helping the Noncompliant Child" (HNC) via weekly sessions and mid-week calls.
  Helping the Noncompliant Child (HNC): HNC is a mastery-based, family-focused, clinic-based treatment for young children aged 3-8 years with problem behavior.
Period: Overall Study
Arm/Group | Helping the NonCompliant Child Treatment
Started | 45
Completed | 10
Not Completed | 35

BASELINE CHARACTERISTICS:
Arm/Group | Helping the NonCompliant Child Treatment
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.83 (1.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 36
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Eyberg Child Behavior Inventory (ECBI) Score-Intensity
Description: The ECBI is a 36 item parent-report scale. For each item, parents rate the intensity of the behavior (0 = never to 7 = always) and whether they consider each behavior to be a problem (0 = no; 1 = yes). Clinically significant symptoms are defined by scores more than 2 standard deviations above the normed mean for the Intensity Subscale (clinical cutoff = 127) and/or Problem Subscale (clinical cutoff = 11) Scales. Intensity scores range from 36 to 252. A mean score decrease indicates a reduction in parent perception of the intensity of the problem behavior.
Time Frame: Baseline, study completion, approximately 10 weeks total
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Helping the NonCompliant Child Treatment
Number analyzed (Participants) | 35
score on a scale | -45.46 [-101.0 to -4.0]

2. Primary Outcome: Change in Eyberg Child Behavior Inventory (ECBI) Score-Problem
Description: The ECBI is a 36 item parent-report scale. For each item, parents rate the intensity of the behavior (0 = never to 7 = always) and whether they consider each behavior to be a problem (0 = no; 1 = yes). Clinically significant symptoms are defined by scores more than 2 standard deviations above the normed mean for the Intensity Subscale (clinical cutoff = 127) and/or Problem Subscale (clinical cutoff = 11) Scales. The number of "yes" responses are counted and averaged. Problem scores range from 0 to 36. A mean score decrease indicates a reduction in parent perception of the number of the problem behaviors.
Time Frame: Baseline, study completion, approximately 10 weeks total
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Helping the NonCompliant Child Treatment
Number analyzed (Participants) | 35
score on a scale | -9.37 [-24.0 to 4.0]

3. Secondary Outcome: Change in Difficulties With Emotion Regulation Scale (DERS) Score
Description: The Difficulties in Emotion Regulation Scale (DERS) will be used as the measure of caregiver's emotion dysregulation. The 36-item DERS yields a composite total score as well as scores for the following subscales: 1) Nonacceptance Subscale, non-acceptance of negative emotions; 2) Goal Subscale, difficulties in engaging in goal-directed behaviors when experiencing negative emotions, 3) Impulse Subscale, impulse control difficulties; 4) Strategies Subscale, limited access to emotion regulation strategies; 5) Awareness Subscale, lack of emotional awareness; and 6) Clarity Subscale, lack of emotional clarity. DERS total scores range from 36 to 180. The composite total is reported for this small sample size. A mean score decrease indicates a reduction in parent difficulties with emotion regulation.
Time Frame: Baseline, study completion, approximately 10 weeks total
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Helping the NonCompliant Child Treatment
Number analyzed (Participants) | 35
score on a scale | -1.11 [-39.0 to 82.0]

4. Secondary Outcome: Change in Coping With Children's Negative Emotions Scale Score
Description: The Coping with Children's Negative Emotions Scale (CCNES) assesses the ways that parents cope with their children's distress and negative emotions. Participants use a 7-point Likert scale where 7 indicates high levels of specific parenting behavior (i.e. supportive and non-supportive parenting behavior). Scores are reported condensing 6 categories into 2 broader domains (supportive/non-supportive) with scores ranging from 1 to 21. Assessed at Baseline and end of study. A mean score decrease in non-supportive scores reflects an improvement in parents' non-supportive strategies and a mean score increase in the supportive score indicates improvement in parents' supportive strategies.
Time Frame: Baseline, study completion, approximately 10 weeks total
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Helping the NonCompliant Child Treatment
Number analyzed (Participants) | 35
score on a scale
  Supportive | 0.45 [-2.08 to 1.67]
  Non-Supportive | -1.06 [-5.11 to 1.08]

ADVERSE EVENTS:
Time Frame: From the time of Informed Consent through post assessment visit, an approximate total of 10 weeks.
Arm/Group | Helping the NonCompliant Child Treatment
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT03597789/Prot_SAP_000.pdf